CLINICAL TRIAL: NCT07051850
Title: Observational Study of Quality of Life, Efficacy, and Safety Following Administration of Advanced Immuno-Oncology Agents Versus Conventional Immunotherapies in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Quality of Life and Treatment Outcomes in RRMM Patients Receiving Advanced vs. Conventional Immunotherapies
Status: Recruiting | Type: Observational
Sponsor: Sung-Soo Park (Other)
Collaborators: Eunpyeong St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Sung-Soo Park, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: XC25OIDI0011
Record Dates: First submitted 2025-06-09; First posted 2025-07-04 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma, Relapsed; Multiple Myeloma (MM)
Keywords: Relpased; Refractory; Advanced Immuno-Oncology Agents; Conventional Immunotherapies
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Antibodies, Bispecific; Immunoconjugates; Antibodies, Monoclonal; Proteasome Inhibitors; Immunotherapy, Adoptive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, Bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Advanced Immuno-oncology Therapy Group
  Interventions: Drug: Bispecific antibody; Drug: CAR-T Therapy
- Conventional Immuno-oncology Therapy Group
  Interventions: Drug: Antibody-Drug Conjugate; Drug: Monoclonal antibody; Drug: Proteasome Inhibitor; Drug: IMiD treatment

INTERVENTIONS:
Drug: Bispecific antibody — It uses a dual targeting mechanism to enhance specificity and immune activation. It is an off-the-shelf treatment, and doesn't require a manufacturing process of patient cells.
  Groups: Advanced Immuno-oncology Therapy Group
Drug: Antibody-Drug Conjugate — It is a targeted therapy consisting of a monoclonal antibody linked to a cytotoxic drug. The antibody binds to a specific antigen on cancer cells, delivering the cytotoxic agent directly to the tumor, minimizing systemic toxicity.
  Groups: Conventional Immuno-oncology Therapy Group
Drug: Monoclonal antibody — Monoclonal antibodies are lab-engineered antibodies that target specific antigens expressed on cancer cells. These commonly target CD20 (rituximab or obinutuzumab) to mediate immune destruction.
  Groups: Conventional Immuno-oncology Therapy Group
Drug: Proteasome Inhibitor — It blocks the activity of proteasomes, which role is degrading damaged proteins. This disruption induces apoptosis in cancer cells. Common agents include bortezomib and carfilzomib.
  Groups: Conventional Immuno-oncology Therapy Group
Drug: IMiD treatment — Immune modulatory drugs modulate the immune response by enhancing T-cell and NK cell activty to disrupt tumor progression. Common drugs include lenalidomide and thalidomide.
  Groups: Conventional Immuno-oncology Therapy Group
Drug: CAR-T Therapy — It uses the patient's own T cells, and requires a manufacturing process to modify and expand T cells before infusion. It directly targets B cell specific antigens, such as CD19 or CD20.
  Groups: Advanced Immuno-oncology Therapy Group

SUMMARY:
This is a non-interventional observational study aiming to evaluate the quality of life, efficacy, and safety of advanced immuno-oncology agents versus conventional immuno-oncology therapies in patients with relapsed or refractory multiple myeloma. A total of 174 participants are expected to be enrolled in this study.

The study consists of three parts:

Part 1 is the screening and enrollment phase, during which inclusion and exclusion criteria will be assessed for individuals who have agreed to participate in the study. Eligible participants will be enrolled, and data will be collected on their prioritized treatment value criteria.

Part 2 is the treatment phase, during which participants will receive either conventional immuno-oncology therapy or advanced immuno-oncology agents. Participants will visit the site on Day 1 of each treatment cycle to complete patient-reported outcomes (PROs), and efficacy and safety assessments will be conducted.

Part 3 is the end-of-study visit, during which PROs will again be collected, along with final efficacy and safety assessments.

Additionally, for exploratory purposes, bone marrow and peripheral blood samples will be collected from participants at Seoul St. Mary's Hospital who have consented to sample collection and provision during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 19 years or older.
* Diagnosed with multiple myeloma and have been previously treated with at least one proteasome inhibitor, one immunomodulatory drug, and one monoclonal antibody treatment (i.e., exposed to all three classes of immunotherapy agents).
* Diagnosed with relapsed or refractory multiple myeloma between the IRB approval date and December 2025, and scheduled to start treatment with either advanced immuno-oncology agents or conventional immuno-oncology agents within one month from screening.
* Provided written informed consent after receiving detailed explanation about the study and voluntarily agreed to participate and comply with study requirements.

Exclusion Criteria:

* Those who do not agree to participate in the study.
* Patients diagnosed with plasma cell disorders other than multiple myeloma (e.g., lymphoma, POEMS syndrome).
* Individuals unable to read and understand documents written in Korean.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from Seoul St. Mary hospital and Yeoido St. Mary hospital
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Lfe | From treatment initiation up to 12 months
  Quality of life is assessed using validated patient-reported outcome (PRO) questionnaires at baseline and regular intervals during treatment.

SECONDARY OUTCOMES:
Treatment Efficacy and Survival Outcomes | From treatment initiation up to 12 months
  Treatment Efficacy will be assessed by objective response rate (ORR), progression-free survival (PFS), and overall survival (OS). ORR will be reported as the percentage of participants with complete or partial response per IMWG criteria, based on clinical and imaging assessments. PFS and OS will be measured in months as time-to-event outcomes.
  Survival Outcomes will be evaluated by the number of participants with adverse events (AEs) and serious adverse events (SAEs), graded using CTCAE. Laboratory safety will be assessed by the number of participants with CTCAE-defined lab abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary Hospital, Seocho, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No